CLINICAL TRIAL: NCT00037921
Title: UTI Prophylaxis Using Bacterial Interference Following SCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Darouiche, Rabih - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: B2410R
Record Dates: First submitted 2002-05-24; First posted 2002-05-27 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-05

CONDITIONS: Urinary Tract Infections
Keywords: SCI; UTI
MeSH Terms: conditions — Urinary Tract Infections

ARMS (1):
- 1 (Other)
  Interventions: Procedure: Bacterial colonization

INTERVENTIONS:
Procedure: Bacterial colonization

SUMMARY:
Urinary tract infection (UTI) is the most common infection in patients with SCI and is a major cause of morbidity and mortality in this population. The bladder of patients with SCI, especially those who have indwelling catheters, is often colonized by bacteria that may or may not cause symptoms of UTI. Bacteria that do not cause symptoms are usually considered benign colonizers and are often left untreated because they may afford some protection against symptomatic infection with more harmful bacteria.

We applied the concept of using benign bacteria to prevent symptomatic infection, so-called bacterial interference, by deliberately colonizing the bladder of patients with SCI with a non-pathogenic prototype of Escherichia coli (strain 83972). The preliminary results of our VA-funded study that compared the rates of symptomatic UTI in patients with SCI while colonized with E. coli 83972 vs. historical rates of symptomatic UTI prior to study enrollment indicated that deliberate colonization of the bladder of patients with SCI with E. coli 83972 is safe and very promising as to its ability to prevent symptomatic UTI. However, before this innovative approach of bacterial interference can be successfully applied in the population of patients with SCI, it is essential to: (A) confirm the ultimate efficacy of bacterial interference by conducting a prospective, randomized, placebo-controlled clinical trial (objective #1); and (B) enhance the practicality of applying this innovative approach in SCI patients by delineating the bacterial and host factors that can promote successful colonization with E. coli 83972 (objectives #2-3).

DETAILED DESCRIPTION:
A prospective, randomized, placebo-controlled clinical trial will be conducted. Patients who had sustained SCI >18 months earlier, suffer from neurogenic bladder (require intermittent bladder catheterization, an indwelling suprapubic catheter, or an external collection device), and have a history of frequent symptomatic UTI (> 2 episodes during the preceding year) will be eligible for enrollment. Exclusion criteria will include urolithiasis, indwelling nephrostomy catheter, indwelling transurethral foley catheter, supravesical urinary diversion, vesicoureteral reflux, conditions anticipated to require antibiotic therapy for chronic recurrent extraurogenital infections (e.g. infected decubitus ulcers), uncontrolled diabetes mellitus and immunosuppression. Patients considered unreliable to pursue adequate follow-up and those incapable of giving informed consent will also be excluded. Subjects will discontinue all measures to suppress UTI for at least two weeks prior to entry into the study. All patients will have a complete history and physical examination, serum creatinine, plain X-ray of the abdomen (KUB), and urine culture immediately prior to entry into the study. Renal ultrasound and urodynamic evaluation of the urinary tract will also be obtained upon study entry unless they have been performed during the preceding year.

ELIGIBILITY:
Inclusion Criteria:

SCI UTI

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2001-01; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rabih Darouiche, MD, Principal Investigator — Michael E. DeBakey VA Medical Center (152)
Locations (1):
- Michael E. DeBakey VA Medical Center (152), Houston, Texas, United States